CLINICAL TRIAL: NCT03995329
Title: Acute Effects of a Heat-not-burn Tobacco Product on Pulmonary Function in Healthy Non Smokers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Athanasia Pataka, Assistant Professor of Respiratory Medicine, Aristotle University Of Thessaloniki
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 762.18/06/2019
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Heated Tobacco; Respiratory Function; Tobacco Toxicity
Keywords: pulmonary function; heated tobacco; IQOS
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy non smokers (Other): Healthy non smokers males, aged 18-55years,receiving no medications
  Intervention: the use of an IQOS Examination of pulmonary function, exhaled CO, blood pressure, heart rate and O2 saturation immediatly after IQOS
  Interventions: Other: IQOS

INTERVENTIONS:
Other: IQOS — Acute effects of IQOS on pulmonary function, oxygen saturation, exhaled CO, heart rate and arterial blood pressure.

SUMMARY:
IQOS ("I-Quit-Ordinary-Smoking,") is a type of "heat-not-burn" (HNB) tobacco product. There is evidence of a growing number of young people who try IQOS as a 'safe' alternative of cigarette. The effect of the acute exposure to IQOS smoke on pulmonary function of healthy non smokers has not been studied extensively.

Objectives: Evaluation of the acute effects of IQOS on pulmonary function,exhaled CO, O2 Saturation, arterial pressure and heart rate.

Methods: Healthy non smokers, underwent exhaled CO measurement, spirometry including flows, volumes and diffusion capacity, and measurement of their respiratory resistances at 5, 10 and 20 Hz (R5Hz, R10Hz and R20Hz) with the use of an impulse oscillometry system (IOS) before and after the use of an IQOS. Additionally heart rate and arterial blood pressure were also measured.

DETAILED DESCRIPTION:
All participants underwent pulmonary function tests (PFT) (MasterScreen PFT, Jaeger, Wurzburg, Germany) and total respiratory resistances measurement with an impulse oscillometry system (IOS)( (Viasys Jaeger MasterScreen IOS system).From the basic pulmonary measurements (flows and dynamic lung volumes), Forced Expiratory Volume in 1 second (FEV1), Forced Vital Capacity (FVC), Tiffenau index (FEV1/FVC, FEV1%), Peak Expiratory Flow (PEF), Maximal Expiratory Flow (MEF) at 25%, 50%, and 75% of vital capacity, Functional Residual Capacity (FRC), Total Lung Capacity (TLC), Residual Volume (RV), Diffusion Capacity (DLCO) were measured. Each manoeuvre was repeated for at least three technically acceptable forced expiratory flow curves in order to attain the best results. Respiratory impedance at 5 Hz (Z5Hz) and respiratory resistance at 5, 10, and 20 Hz (R5Hz, R10Hz, and R20Hz, respectively), reactance at 5, 10, and 20 Hz and resonant frequency were assessed with IOS. Heart rate, saturation of O2 (oxymetry) and arterial blood pressure were also measured. Exhaled CO measurement (piCO Smokerlyzer,Bedfont Scientific Ltd, Kent, U.K.) was performed After smoking heated tobacco (IQOS): 5 minutes after smoking IQOS , they repeated again PFTs, IOS, exhaled CO heart rate, saturation of O2 (oximetry) and arterial blood pressure measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male non smokers,
2. Age 18-55 years
3. receiving no medications
4. no co morbidity -

Exclusion Criteria:

1. aged <18 years
2. smokers or ex-smokers
3. receiving any medications
4. any co morbidity -

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second | immediately (max 5 min)
  Pulmonary function tests (PFT) prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in:Forced Expiratory Volume in 1 second (FEV1), (liters)
Forced Vital Capacity | immediatly (max 5 min)
  Pulmonary function tests (PFT) prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in:Forced Vital Capacity (FVC), (liters)
Tiffenau index | immediately (max 5 min)
  Pulmonary function tests (PFT) prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in:
  Tiffenau index (FEV1/FVC, FEV1%)
Peak Expiratory Flow | immediately (max 5 min)
  Pulmonary function tests (PFT) prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in: Peak Expiratory Flow (PEF), (liters/second )
Functional Residual Capacity (FRC) | immediately (max 5 min)
  Pulmonary function tests (PFT) prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in:Functional Residual Capacity (FRC), (liters)
Total Lung Capacity (TLC) | immediately (max 5 min)
  Pulmonary function tests (PFT) prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in: Total Lung Capacity (TLC), (liters)
Residual Volume (RV) | immediately (max 5 min)
  Pulmonary function tests (PFT) prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in: Residual Volume (RV), (liters)
Diffusion Capacity (DLCO) | immediately (max 5 min)
  Pulmonary function tests (PFT) prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in: Diffusion Capacity (DLCO) ((mmol/min/kPa)
Respiratory impedance | immediately (max 5 min)
  Total respiratory resistances measurement with an impulse oscillometry system (IOS)( (Viasys Jaeger MasterScreen IOS system) prior to smoking heated tobacco IQOS and 5 minutes after smoking IQOS were performed. The changes in: Respiratory impedance at 5 Hz (Z5Hz) (kPa/L/sec) were assessed
Total respiratory resistances | immediately (max 5 min)
  Total respiratory resistances measurement with an impulse oscillometry system (IOS)( (Viasys Jaeger MasterScreen IOS system) prior to smoking heated tobacco IQOS and 5 minutes after smoking IQOS were performed. The changes in: respiratory resistance at 5 (R5Hz),10 Hz (R10Hz),20 Hz (R20Hz) (kPa/L/sec) were assessed
Arterial Blood Pressure | immediately (max 5 min)
  Arterial Blood Pressure prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in Arterial Blood Pressure were measured (mmHg)
Oxygen Saturation | immediately (max 5 min)
  Oxygen Saturation prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in Oxygen Saturation were measured by oximetry
Heart rate | immediately (max 5 min)
  Heart rate prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in Heart rate were measured by oximetry
Exhaled CO | immediately (max 5 min)
  Exhaled CO prior to smoking heated tobacco IQOS and 5 minutes after IQOS. The changes in Exhaled CO were measured by (piCO Smokerlyzer) (ppm)

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - G Papanicolaou Hospital, Thessaloniki, Thessaloniki
  - Respiratory Failure Unit, G Papanikolaou Hospital, Aristotle Unioversity of Thessaloniki, Thessaloniki

IPD SHARING:
Plan to Share IPD: No